CLINICAL TRIAL: NCT04579068
Title: Alcohol Awareness Peer Leaders (AAPL): A Multidisciplinary, Culturally Based Training Program for Underserved Minority Health Professional Students to Increase Alcohol Screening and Intervention
Brief Title: Decreasing Alcohol Use Through Student Peer Leaders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not funded
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AAPLCDU
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Alcohol Abuse; Alcohol Drinking; Alcohol Use Disorder; Alcohol Problem
Keywords: alcohol
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Alcohol-Related Disorders | interventions — Mass Screening; Ethanol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening and Brief Intervention of Problematic Alcohol Use (Experimental): We plan to test the feasibility and effectiveness of the delivery of the peer-based SBIRT using the RAPS4-QF screening tool with CDU students. Furthermore, we will compare delivery by AAPLs' race/ethnicity, drinking status (abstainer vs. non-abstainer), and adverse life experiences. Following the screening by AAPLs, we expect a 30% detection of problematic alcohol use (i.e. high episodic drinking [HED] or AUD) and at-risk alcohol use. Participants that screen positive will receive brief motivational interviewing and referral to treatment and will be contacted 6 months following the SBIRT to assess their drinking behaviors. We expect that participants will decrease their alcohol consumption or drinking risk at the 6-month follow up.
  Interventions: Behavioral: Screening and Brief Intervention of Problematic Alcohol Use

INTERVENTIONS:
Behavioral: Screening and Brief Intervention of Problematic Alcohol Use — Provide/enhance knowledge, screening and detection, modify attitudes, motivate and provide skills and resources to reduce alcohol related risk and consumption.

SUMMARY:
Problematic alcohol use can lead to worse social and health related consequences for underserved minorities, requiring urgent intervention. By training underserved minority health professional students, this proposed project will develop and test the feasibility of an innovative and culturally tailored intervention for adults studying at a minority institution, with specific focus on alcohol screening, brief intervention, and referral of treatment (SBIRT). This proposal is expected to have a positive impact on alcohol reduction and prevention for minority communities

DETAILED DESCRIPTION:
Problematic alcohol use, including alcohol use disorders (AUD) and high episodic drinking (HED), remains a public health crisis among college students, particularly those from underserved minority groups. Less likely to disclose alcohol use, underserved minority college students participate in riskier drinking, attributed to multiple social factors, including racial/ethnic discrimination, financial strain, and neighborhood disadvantage. Faced with worse alcohol health-related consequences, effective interventions to reduce alcohol use among this population is critically needed. To reduce alcohol-related health disparities, the investigators aim to develop a public health-based, comprehensive program (Alcohol Awareness Peer Leaders) that will train underserved minority non-traditional health professional students to conduct alcohol screening, brief intervention, and referral to treatment (SBIRT) by using a culturally sensitive approach and screening tool (Rapid Alcohol Problems Screen - RAPS4-QF). By utilizing a culturally adapted SBIRT curriculum, AAPLs will be able to deliver alcohol education and messaging to motivate alcohol risk reduction and decrease in consumption for non-traditional college students studying at a predominantly minority academic institution in an underserved area. The Andersen Healthcare Utilization Model will be utilized to guide this intervention. This theoretically and culturally tailored proposed project is evidence-informed and promising for underserved minority college students and will be advanced through the following three aims: 1) Using an explanatory-sequential mixed methods design, examine a) alcohol consumption and HED patterns, b) attitudes toward alcohol use, c) social and environmental factors, and d) alcohol-related consequences among minority health professional students, 2) Through training of minority health professional students as Alcohol Awareness Peer Leaders (AAPLs), assess the acceptability and relevance of a peer-based SBIRT that was culturally-tailored based on Aim 1 findings, and 3) To compare the feasibility and effectiveness of delivering a culturally-tailored SBIRT using RAPS4-QF by AAPLs by race/ethnicity, drinking status (abstainer vs. drinker), and adverse life experiences. These outcomes will result in the training of 208 underserved minority AAPLs who will conduct culturally competent and evidence-based alcohol screening, brief intervention, and treatment referral for over 2000 students. The result of this innovative proposal will produce future healthcare professionals who will be a valuable community resource for underserved areas as they can continue to decrease alcohol health disparities for underrepresented minority populations, inducing sustainability.

ELIGIBILITY:
Inclusion Criteria:

* enrolled student at CDU
* age 18 or older
* Speak and understand English

Exclusion Criteria:

* not enrolled as a student at CDU
* Under the age of 18
* Unable to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-21 (Estimated); Primary Completion 2026-08-21 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Detection of problematic alcohol use (i.e. HED or AUD) and at-risk alcohol use Using the RAPS4-QF Instrument | 15 minutes
  Following the RAPS4-QF screening by AAPL, we anticipate that we will detect a 30% detection of problematic alcohol use (i.e. HED or AUD) and at-risk alcohol use.
Detection of problematic alcohol use (i.e. HED or AUD) and at-risk alcohol use based on adverse life experiences Using the RAPS4-QF Instrument | 15 minutes
  Following the RAPS4-QF screening by AAPL, we anticipate that AAPLs with adverse life experiences will have a 40% detection rate of problematic alcohol use (i.e. HED or AUD) and at-risk alcohol use.
Detection of problematic alcohol use (i.e. HED or AUD) and at-risk alcohol use based on Race/Ethnicity Using the RAPS4-QF Instrument | 15 minutes
  Following the RAPS4-QF screening by AAPL, we anticipate that AAPLs with matching race/ethnicity will have a 30% detection rate of problematic alcohol use (i.e. HED or AUD) and at-risk alcohol use.
Detection of problematic alcohol use (i.e. HED or AUD) and at-risk alcohol use based on drinking status Using the RAPS4-QF Instrument | 15 minutes
  Following the RAPS4-QF screening by AAPL, we anticipate that AAPLs that are alcohol non-abstainers will have a 30% detection rate of problematic alcohol use (i.e. HED or AUD) and at-risk alcohol use.
Percentage of Participants Achieving Decreased Levels of Alcohol Risk Using the SBIRT Intervention | Intervention: 15 minutes; Follow-up Point: 6 months post-intervention
  By comparison of pre-, post- intervention, and six-months follow-up data, we anticipate the following compared to baseline: a 30% change in alcohol risk.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Cobb, PhD, Principal Investigator — Charles R. Drew University of Medicine & Science